CLINICAL TRIAL: NCT02325986
Title: Concurrent Radiotherapy and Weekly Chemotherapy of 5-fluorouracil and Cisplatin for Postoperative Locoregional Recurrence of Oesophageal Squamous Cell Carcinoma
Brief Title: Concurrent Radiotherapy and Weekly Chemotherapy of PF for Postoperative Locoregional Recurrence of Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhu Yujia, Attending physicion, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GD-B2014157
Record Dates: First submitted 2014-12-16; First posted 2014-12-25 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: radiotherapy; esophageal carcinoma; chemotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms | interventions — Fluorouracil; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Weekly PF with radiation (Experimental): 4 cycles of weekly cisplatin and fluorouracil (cisplatin 25mg/m2 on day 1, fluorouracil 1176mg/m2 on day 1-3, repeated weekly for 4 weeks) concurrently with Intensity-modulated radiation therapy (60Gy/28fr).
  Interventions: Drug: fluorouracil; Drug: Cisplatin; Radiation: Intensity-modulated radiation therapy

INTERVENTIONS:
Drug: fluorouracil — cisplatin 25mg/m2 on day 1, fluorouracil 1176mg/m2 on day 1-3，repeated weekly for 4 weeks concurrently with IMRT radiotherapy (60Gy/28fr)
  Other Names: 5-FU
Drug: Cisplatin — cisplatin 25mg/m2 on day 1, fluorouracil 1176mg/m2 on day 1-3，repeated weekly for 4 weeks concurrently with IMRT radiotherapy (60Gy/28fr)
Radiation: Intensity-modulated radiation therapy — cisplatin 25mg/m2 on day 1, fluorouracil 1176mg/m2 on day 1-3，repeated weekly for 4 weeks concurrently with IMRT radiotherapy (60Gy/28fr)
  Other Names: IMRT

SUMMARY:
The purpose of this study is to evaluate the efficacy and toxicity of radiotherapy concurrently with weekly chemotherapy of 5-FU and cisplatin in patients with postoperative locoregional recurrence of esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
The most optimal management for postoperative locoregional recurrence of oesophageal squamous cell carcinoma is still controversial. Several studies have reported the feasibility and efficacy of concurrent chemoradiotherapy (CCRT), mostly with three-weekly or four-weekly schedule of chemotherapy. However, treatment compliance was not quite satisfactory, probably due to treatment-related toxicities. Since CCRT with weekly chemotherapy regimens have demonstrated a favorable toxicity profile as well as promising survival in certain types of cancer, the investigators aimed to evaluate the efficacy and toxicity of radiotherapy concurrently with weekly chemotherapy with 5-fluorouracil (5-FU) and cisplatin for patients with postoperative locoregional recurrence of oesophageal squamous cell carcinoma in the investigators center.The prescribed dose of radiotherapy is generally 60Gy/28fr to tumor and 50Gy/28fr to the clinical target volume.The concomitant chemotherapy is cisplatin 25mg/m2 on day 1, 5-FU 1176mg/m2 on day 1-3, repeated weekly for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. R0 resection for primary esophageal squamous cell carcinoma with two-incision esophagectomy (Ivor Lewis approach)25 or three-incision (right thoracotomy, midline laparotomy and left cervical incisions) esophagectomy with cervical esophagogastric anastomosis.
2. Absence of previous thoracic radiotherapy.
3. Cervical and/or thoracic postoperative recurrence (biopsy proven or positron emission tomography/computed tomography (PET/CT) proven or follow-up computed tomography (CT) showed progression of disease).
4. Absence of distant metastasis at recurrence.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2

Exclusion Criteria:

1. Younger than 18 or older than 70 years of age.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 3 or above
3. Other cancer history.
4. Serious cardiac, liver, or pulmonary disease.
5. Previous radiotherapy history

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
overall response rate | within 8 weeks after the treatment(plus or minus 5 days)
  RECIST (Response Evaluation Criteria in Solid Tumors) was used to determine the tumor response. Tumor response was evaluated by CT 8 weeks after chemoradiotherapy.

SECONDARY OUTCOMES:
safety: Toxicity was graded according to the Common Terminology Criteria for Adverse Events (CTCAE v3.0). | up to 3 years
  A 3 years follow-up from the enrollment or to the date of death from any cause or date of lost follow-up
overall survival | up to 3 years
  A 3 years follow-up from the enrollment or to the date of death from any cause or date of lost follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Yujia Zhu, MD, Principal Investigator — Department of Radiation Oncology, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, P.R. China
Locations (1):
- SYSU Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Rice TW, Rusch VW, Apperson-Hansen C, Allen MS, Chen LQ, Hunter JG, Kesler KA, Law S, Lerut TE, Reed CE, Salo JA, Scott WJ, Swisher SG, Watson TJ, Blackstone EH. Worldwide esophageal cancer collaboration. Dis Esophagus. 2009;22(1):1-8. doi: 10.1111/j.1442-2050.2008.00901.x. PMID 19196264
- [Background] Kato H, Miyazaki T, Nakajima M, Sohda M, Fukai Y, Masuda N, Fukuchi M, Manda R, Tsukada K, Kuwano H. Prediction of hematogenous recurrence in patients with esophageal carcinoma. Jpn J Thorac Cardiovasc Surg. 2003 Nov;51(11):599-608. doi: 10.1007/BF02736700. PMID 14650590
- [Background] Nakamura T, Ota M, Narumiya K, Sato T, Ohki T, Yamamoto M, Mitsuhashi N. Multimodal treatment for lymph node recurrence of esophageal carcinoma after curative resection. Ann Surg Oncol. 2008 Sep;15(9):2451-7. doi: 10.1245/s10434-008-0016-x. Epub 2008 Jul 1. PMID 18592318
- [Background] Shioyama Y, Nakamura K, Ohga S, Nomoto S, Sasaki T, Yamaguchi T, Toba T, Yoshitake T, Terashima H, Honda H. Radiation therapy for recurrent esophageal cancer after surgery: clinical results and prognostic factors. Jpn J Clin Oncol. 2007 Dec;37(12):918-23. doi: 10.1093/jjco/hym138. PMID 18211982
- [Background] Kobayashi R, Yamashita H, Okuma K, Shiraishi K, Ohtomo K, Nakagawa K. Salvage radiation therapy and chemoradiation therapy for postoperative locoregional recurrence of esophageal cancer. Dis Esophagus. 2014 Jan;27(1):72-8. doi: 10.1111/dote.12068. Epub 2013 Apr 2. PMID 23551708
- [Result] Yuan G, Wu L, Huang M, Li N, An J. A phase II study of concurrent chemo-radiotherapy with weekly nedaplatin in advanced squamous cell carcinoma of the uterine cervix. Radiat Oncol. 2014 Feb 18;9:55. doi: 10.1186/1748-717X-9-55. PMID 24533532
- [Result] Nakagawa S, Kanda T, Kosugi S, Ohashi M, Suzuki T, Hatakeyama K. Recurrence pattern of squamous cell carcinoma of the thoracic esophagus after extended radical esophagectomy with three-field lymphadenectomy. J Am Coll Surg. 2004 Feb;198(2):205-11. doi: 10.1016/j.jamcollsurg.2003.10.005. PMID 14759776
- [Result] Stahl M, Stuschke M, Lehmann N, Meyer HJ, Walz MK, Seeber S, Klump B, Budach W, Teichmann R, Schmitt M, Schmitt G, Franke C, Wilke H. Chemoradiation with and without surgery in patients with locally advanced squamous cell carcinoma of the esophagus. J Clin Oncol. 2005 Apr 1;23(10):2310-7. doi: 10.1200/JCO.2005.00.034. PMID 15800321
- [Result] Bao Y, Liu S, Zhou Q, Cai P, Anfossi S, Li Q, Hu Y, Liu M, Fu J, Rong T, Li Q, Liu H. Three-dimensional conformal radiotherapy with concurrent chemotherapy for postoperative recurrence of esophageal squamous cell carcinoma: clinical efficacy and failure pattern. Radiat Oncol. 2013 Oct 18;8:241. doi: 10.1186/1748-717X-8-241. PMID 24139225
- [Result] Jingu K, Nemoto K, Matsushita H, Takahashi C, Ogawa Y, Sugawara T, Nakata E, Takai Y, Yamada S. Results of radiation therapy combined with nedaplatin (cis-diammine-glycoplatinum) and 5-fluorouracil for postoperative locoregional recurrent esophageal cancer. BMC Cancer. 2006 Mar 4;6:50. doi: 10.1186/1471-2407-6-50. PMID 16515704
- [Result] Ma DY, Tan BX, Liu M, Li XF, Zhou YQ, Lu Y. Concurrent three-dimensional conformal radiotherapy and chemotherapy for postoperative recurrence of mediastinal lymph node metastases in patients with esophageal squamous cell carcinoma: a phase 2 single-institution study. Radiat Oncol. 2014 Jan 19;9:28. doi: 10.1186/1748-717X-9-28. PMID 24438695